CLINICAL TRIAL: NCT00764894
Title: Post-Market Study of the Foundation Knee System
Brief Title: Foundation Knee Study - Retrospective
Status: Terminated | Type: Observational
Why Stopped: Enrollment and data collection insufficient to continue study.
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Other Study IDs: PS - 701
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Inflammatory Tissue Disorders; Arthritis Secondary to Other Diseases; Avascular Necrosis of the Femoral Condyles
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Foundation Knee: Retrospective data collection on 510(k) approved device
  Interventions: Device: Foundation Knee

INTERVENTIONS:
Device: Foundation Knee — Subjects with degenerative joint disease (DJD), osteoarthritis or rheumatoid arthritis who received a primary Foundation Knee replacement and is willing to participate in the study.

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the Encore Foundation Knee System in a group of 200 patients for whom data has already been collected.

ELIGIBILITY:
Inclusion Criteria:

* Have knee joint disease related to one or more of the following

  * osteoarthritis
  * post-traumatic arthritis
  * inflammatory tissue disorders
  * arthritis secondary to other diseases
  * Avascular necrosis of the femoral condyles;
* Skeletal maturity
* Less than 70 on the Knee Society Score (rating score)
* Sufficient bone stock, as judged by radiographs, to support primary knee implant
* Sufficient collateral ligaments to support the device, as judged by physician during stability testing (varus/valgus and flexion/extension) and less than 45 degree varus/valgus deformity and/or 90 degree flexion contracture
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures
* Patient is not pregnant
* No infection present
* No known materials sensitivity

Exclusion Criteria:

* Skeletal immaturity
* Greater than or equal to 70 on preoperative Knee Society Score (Rating Score)
* Post-patellectomy
* Insufficient bone quality which may affect implant stability
* Insufficient collateral ligaments, as judged by the physician. Greater than 45 degree varus/valgus deformity and/or 90 degree flexion contracture.
* Neurological conditions that might hinder patient's ability to follow study procedures (i.e., any that restrict physical activities such as Parkinson's Disease, Multiple Sclerosis, previous stroke which affects lower extremity)
* Mental conditions that may interfere with ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the patient cannot understand the informed consent process, global dementia, prior strokes that interfere with the patient's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Prisoners
* Conditions that place excessive demand on the implant (i.e. Charcot's joints, muscle deficiencies, refusal to modify postoperative physical activities, skeletal immaturity)
* Patient is pregnant
* Infection present
* Materials sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who meet the indications for use of the Foundation Knee device AND who meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The use and efficacy of the Encore Foundation Knee System | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Omar Hussamy, M.D., Principal Investigator — Hussamy Orthopedics
Locations (1):
- Hussamy Orthopedics, Vero Beach, Florida, United States

REFERENCES:
- See also: Sponsor Company home page — http://www.djosurgical.com